CLINICAL TRIAL: NCT02246751
Title: Effect of Targeted Training on Sensorimotor Control of Trunk Posture
Brief Title: Case Series_Targeted Training for Trunk Control Cerebral Palsy
Acronym: CP_TT_UHart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hartford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP_TT_2014
Record Dates: First submitted 2014-09-16; First posted 2014-09-23 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Cerebral Palsy
Keywords: postural control; Targeted Training; cerebral palsy; sensorimotor control; trunk segments
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single subject design case series (Experimental): Targeted Training for trunk control, 5-6 days a week for 9 months, minimum of 20 minutes per day.
  Interventions: Device: Targeted Training for trunk control

INTERVENTIONS:
Device: Targeted Training for trunk control — Orthotics Research and Locomotor Research Unit (ORLAU) standers will be custom fit to help the child train at the segmental level of the trunk where they begin to lose control of posture. The typical course of treatment involves loaning the customized equipment to each family for use in their home or in their child's educational setting. Training occurs once daily usually for 30-45 minutes. This is done 5 or 6 days per week. Training programs typically involve playing with balls or balloons or video games that motivate the child to hold the head erect and to wave the arms and hands and move the upper body. The researchers evaluate children every 8 weeks and adjust the stander to lower levels of support as the child gains control.
  Other Names: Segmental training for trunk control

SUMMARY:
Little is known about how children with cerebral palsy (CP) use their sensory systems (touch, sense of body position, balance organs in the inner ear, vision) to help them achieve trunk control for independent sitting. If a child with CP does not achieve trunk control by 4 years of age their prognosis for motor skill development including walking is poor. Clinical researchers at The Movement Centre in Oswestry, England have developed a method called Targeted Training in which children train trunk control in small segments from the top down using a custom fit training device. This study aims to examine how children with moderate to severe CP use sensory information for trunk control before, during and after a program of Targeted Training.

DETAILED DESCRIPTION:
One of the major challenges of motor control is to understand how the central nervous system controls the degrees of freedom of the body. This is particularly evident in cerebral palsy (CP), which is the most prevalent chronic childhood motor disability and is one of the most disabling and costly chronic disorders of children and adults. Deficits in postural control and sensorimotor integration are hallmarks of CP. Although postural control of the trunk for independent sitting creates the foundation for all other motor tasks, surprisingly little is known about how children with CP use sensory input to guide their development of upright control (which occurs in typically developing infants by 8 months of age). This lack of knowledge limits our ability to effectively assess and treat children with neuromotor deficits in trunk control.

The objectives of this project are to identify sensory reliance and sensory re-weighting in a study of children with moderate-to-severe CP (4-12 years of age) before and after Targeted Training for Trunk Control. A novel trunk support device will enable testing of participants who lack (or are still developing) stable sitting. In experiments, kinematics of the head and trunk will be measured. Sensory reliance and re-weighting will be identified from postural trunk responses to sensory conflict stimuli consisting of tilts of a visual surround and/or tilts of a surface which participants sit upon. Generally, participants with a high reliance on vestibular feedback will remain upright with respect to gravity during all tests; whereas a high reliance on cutaneous or visual feedback will produce trunk sway away from upright and toward the surface or visual surround tilt, respectively. To tease apart biomechanical, physical, and neurological contributions to trunk sway, sensorimotor integration modeling will be used to complement data interpretation.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy
* age 2-12 years
* Gross Motor Function Classification System (GMFCS) Level III, IV or V

Exclusion Criteria:

* spinal fixation
* fixed scoliosis
* uncontrolled seizures

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change in sensory motor processes | 9 months and 1 and 3 months post training
  Change in sensory motor processes as evidenced by kinematic measures during sitting balance perturbation tasks.

SECONDARY OUTCOMES:
Change in gross motor functional skills (e.g. sitting, crawling, standing) | 9 months and 1 & 3 months post training
  The Gross Motor Function Measure (GMFM 66) is a standardized test of gross motor function that has been validated for children with cerebral palsy
Segmental Assessment of Trunk Control | 2, 4, 6, 8 and 9 months and 1 & 3 months post training
  Change in the trunk segment where static, active or reactive control is lost.

OTHER OUTCOMES:
Participation and Environment Measure for Children and Youth (CY) or Young Children (YC) (PEM-CY for children 5-12 years of age, or YC-PEM for children 2-5 years) | 9 months and 3 months post training
  The PEM-CY and YC-PEM are parent response questionnaires that measure participation frequency, extent of involvement and desire for change in sets of activities typical for the home, school or community.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Saavedra, MS, PT, PhD, Principal Investigator — University of Hartford; Adam Goodworth, MS, PhD, Principal Investigator — University of Hartford
Locations (1):
- Pediatric Balance Laboratory; University of Hartford;, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodworth AD, Peterka RJ. Sensorimotor integration for multisegmental frontal plane balance control in humans. J Neurophysiol. 2012 Jan;107(1):12-28. doi: 10.1152/jn.00670.2010. Epub 2011 Sep 21. PMID 21940611
- [Background] Goodworth AD, Peterka RJ. Contribution of sensorimotor integration to spinal stabilization in humans. J Neurophysiol. 2009 Jul;102(1):496-512. doi: 10.1152/jn.00118.2009. Epub 2009 Apr 29. PMID 19403751
- [Background] Saavedra SL, van Donkelaar P, Woollacott MH. Learning about gravity: segmental assessment of upright control as infants develop independent sitting. J Neurophysiol. 2012 Oct;108(8):2215-29. doi: 10.1152/jn.01193.2011. Epub 2012 Jul 25. PMID 22832568
- [Background] Butler PB, Saavedra S, Sofranac M, Jarvis SE, Woollacott MH. Refinement, reliability, and validity of the segmental assessment of trunk control. Pediatr Phys Ther. 2010 Fall;22(3):246-57. doi: 10.1097/PEP.0b013e3181e69490. PMID 20699770